CLINICAL TRIAL: NCT00183651
Title: Assessment and Treatment of Parasuicidal Patients
Brief Title: Treatment of Suicidal Women With Borderline Personality Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Marsha Linehan, Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01MH034486 (NIH); R01MH034486 (NIH)
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2012-02-02 (Estimated); Status verified 2012-01

CONDITIONS: Borderline Personality Disorder; Suicide
Keywords: Suicide; Women; Emotions; Psychotherapy, Group
MeSH Terms: conditions — Borderline Personality Disorder; Suicide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- S-DBT (Experimental): Participants receive standard dialectical behavior therapy
  Interventions: Behavioral: Standard dialectical behavior therapy (SDBT)
- DBT-I (Active Comparator): Participants receive individual dialectical behavior therapy plus activities group
  Interventions: Behavioral: Individual DBT with no DBT group sessions (DBT-I)
- DBT-S (Active Comparator): Participants receive dialectical behavior therapy group skills plus case management
  Interventions: Behavioral: Group Skills DBT with no DBT individual sessions (DBT-S)

INTERVENTIONS:
Behavioral: Standard dialectical behavior therapy (SDBT) — Standard DBT includes: 1) individual DBT therapy (1 hour per week), 2) DBT group skills training (2.5 hours per week), 3) telephone consultation (as needed), and 4) therapist consultation team (1 hour per week).
  Other Names: DBT, SDBT
  Arms: S-DBT
Behavioral: Individual DBT with no DBT group sessions (DBT-I) — Individual DBT (DBT-I) is 1 hour per week of individual therapy and 2.5 hours per week with the psychosocial activities group.
  Other Names: DBT, DBT-I
  Arms: DBT-I
Behavioral: Group Skills DBT with no DBT individual sessions (DBT-S) — DBT group skills training is 2.5 hours per week and includes individual case management.
  Other Names: DBT, DBT-S
  Arms: DBT-S

SUMMARY:
This study is a component analysis of dialectical behavior therapy (DBT) to determine the importance of DBT skills training and DBT individual therapy in treating suicidal women with borderline personality disorder.

DETAILED DESCRIPTION:
People with borderline personality disorder have limited behavioral skills and react abnormally to emotional stimulation. Standard dialectical behavior therapy (SDBT) has been shown to be an effective treatment for borderline personality disorder. This treatment combines weekly group sessions, at which patients learn new ways of dealing with their emotions, with weekly individual sessions with a therapist to discuss their emotions. The study compares SDBT to both individual DBT with no skills training and DBT skills training with no individual therapy. The study will determine whether efficacy of standard DBT is reduced when either DBT skills training or individual DBT therapy is removed.

Participants are randomly assigned to receive 1 year of SDBT, DBT with group sessions but no individual sessions, and DBT with individual sessions with no group sessions. Participants are monitored for 1 year after completing their assigned therapy. Throughout the 1-year study and during the 1-year follow-up period, self-report scales and questionnaires are used to assess participants every 4 months. These scales and questionnaires measure participants' suicidal thoughts and attempts, treatment compliance, emotional coping skills, social functioning, and overall well-being.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of BPD
* At least one suicide attempt in the year prior to study entry AND at least one intentional self-injury within the 8 weeks prior to study entry
* Willing and able to comply with all study requirements

Exclusion Criteria:

* IQ less than 70
* Life-threatening anorexia
* Street homelessness with no contact information
* Admittance to a hospital with no expectation of discharge within 3 weeks prior to study entry OR sentenced to a jail or prison term that will last for more than 3 weeks
* Ordered by the court to receive psychological treatment
* Meet DSM-IV criteria for schizophrenia, bipolar disorder, or seizure disorder
* Medical conditions other than BPD that may interfere with the study

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 99 (Actual)
Dates: Start 2004-04; Primary Completion 2008-09 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Suicidal thoughts or attempts | Measured at Year 2

SECONDARY OUTCOMES:
Coping skills | Measured at Year 2

CONTACTS AND LOCATIONS:
Overall Officials: Marsha M. Linehan, PhD, Principal Investigator — Department of Psychology, University of Washington
Locations (1):
- University of Washington, Department of Psychology, Behavior Research and Therapy Clinics, Seattle, Washington, United States

REFERENCES:
- [Background] Linehan MM, Armstrong HE, Suarez A, Allmon D, Heard HL. Cognitive-behavioral treatment of chronically parasuicidal borderline patients. Arch Gen Psychiatry. 1991 Dec;48(12):1060-4. doi: 10.1001/archpsyc.1991.01810360024003. PMID 1845222
- [Background] Linehan MM, Tutek DA, Heard HL, Armstrong HE. Interpersonal outcome of cognitive behavioral treatment for chronically suicidal borderline patients. Am J Psychiatry. 1994 Dec;151(12):1771-6. doi: 10.1176/ajp.151.12.1771. PMID 7977884
- [Background] Linehan MM, Dimeff LA, Reynolds SK, Comtois KA, Welch SS, Heagerty P, Kivlahan DR. Dialectical behavior therapy versus comprehensive validation therapy plus 12-step for the treatment of opioid dependent women meeting criteria for borderline personality disorder. Drug Alcohol Depend. 2002 Jun 1;67(1):13-26. doi: 10.1016/s0376-8716(02)00011-x. PMID 12062776
- [Background] Swenson CR, Sanderson C, Dulit RA, Linehan MM. The application of dialectical behavior therapy for patients with borderline personality disorder on inpatient units. Psychiatr Q. 2001 Winter;72(4):307-24. doi: 10.1023/a:1010337231127. PMID 11525079
- [Background] Linehan MM, Schmidt H 3rd, Dimeff LA, Craft JC, Kanter J, Comtois KA. Dialectical behavior therapy for patients with borderline personality disorder and drug-dependence. Am J Addict. 1999 Fall;8(4):279-92. doi: 10.1080/105504999305686. PMID 10598211
- [Background] Verheul R, Van Den Bosch LM, Koeter MW, De Ridder MA, Stijnen T, Van Den Brink W. Dialectical behaviour therapy for women with borderline personality disorder: 12-month, randomised clinical trial in The Netherlands. Br J Psychiatry. 2003 Feb;182:135-40. doi: 10.1192/bjp.182.2.135. PMID 12562741
- [Background] Bohus M, Haaf B, Stiglmayr C, Pohl U, Bohme R, Linehan M. Evaluation of inpatient dialectical-behavioral therapy for borderline personality disorder--a prospective study. Behav Res Ther. 2000 Sep;38(9):875-87. doi: 10.1016/s0005-7967(99)00103-5. PMID 10957822
- [Background] Koons, Cedar R; Robins, Clive J; Tweed, J. Lindsey; Lynch, Thomas R; Gonzalez, Alicia M; Morse, Jennifer Q; Bishop, G. Kay; Butterfield, Marian I; Bastian, Lori A. Efficacy of dialectical behavior therapy in women veterans with borderline personality disorder. Behavior Therapy. Vol 32(2) Spr 2001, 371-390
- [Derived] Witt KG, Hetrick SE, Rajaram G, Hazell P, Taylor Salisbury TL, Townsend E, Hawton K. Psychosocial interventions for self-harm in adults. Cochrane Database Syst Rev. 2021 Apr 22;4(4):CD013668. doi: 10.1002/14651858.CD013668.pub2. PMID 33884617
- [Derived] Storebo OJ, Stoffers-Winterling JM, Vollm BA, Kongerslev MT, Mattivi JT, Jorgensen MS, Faltinsen E, Todorovac A, Sales CP, Callesen HE, Lieb K, Simonsen E. Psychological therapies for people with borderline personality disorder. Cochrane Database Syst Rev. 2020 May 4;5(5):CD012955. doi: 10.1002/14651858.CD012955.pub2. PMID 32368793
- [Derived] Linehan MM, Korslund KE, Harned MS, Gallop RJ, Lungu A, Neacsiu AD, McDavid J, Comtois KA, Murray-Gregory AM. Dialectical behavior therapy for high suicide risk in individuals with borderline personality disorder: a randomized clinical trial and component analysis. JAMA Psychiatry. 2015 May;72(5):475-82. doi: 10.1001/jamapsychiatry.2014.3039. PMID 25806661
- See also: Click here for more information about the Behavioral Research and Therapy Clinics at the University of Washington — http://depts.washington.edu/brtc/